CLINICAL TRIAL: NCT00767208
Title: Comparison of Postprandial Metabolic Responses Between Type 2 Diabetic and Healthy Overweight Subjects
Brief Title: Diabetes and Metabolic Postprandial Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Collaborators: LESAFFRE SA (Unknown)
Responsible Party: Pr Martine Laville, CENTRE DE RECHERCHE EN NUTRITION HUMAINE RHONE ALPES
Model: Parallel | Masking: Single
Other Study IDs: CRNHRA-06-002
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes; Overweight
Keywords: type 2 diabetic subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- type 2 diabetic subjects (Experimental)
  Interventions: Other: oral glucose load
- overweight healthy subjects (Experimental)
  Interventions: Other: oral glucose load

INTERVENTIONS:
Other: oral glucose load — oral ingestion of 13C labeled glucose

SUMMARY:
The aim of this trial was to compare postprandial metabolic response to glucose load in healthy overweight and type 2 diabetic subjects, by using glycemia, insulinemia, lipid profile, nutrient oxidation follow-up. Stable isotopes of glucose were used to assess postprandial total,exogenous and endogenous glucose kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese volunteers
* Healthy for one group nd type 2 diabetic for the second group
* Age between 30 and 65 years old
* Total cholesterol < or = 7 mmol/l and triglycerides < or = 4 mmol/l
* For diabetic group: treated by metformin and/or sulfonylurea and/or thiazolidinedione and HbA1c < 6%
* Stable weight over last 3 months
* Informed consent

Exclusion Criteria:

* No compliant subjects
* Participation in an other trial 2 months before starting this one
* Ward of court or under guardianship (sheltered adults)
* Person deprived of freedom by judicial or administrative decision
* Type 1 diabetes and type 2 diabetes treated bu insulin or acarbose
* Existence of a previously diagnosed pathology (other than type 2 diabetes)
* Previous gastro-intestinal pathology
* Treated by corticoids, anorexigens, weight loss medicines
* Alcoholism or severe tobacco consumption

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Apparition of exogenous glucose in plasma in the postprandial phase and its effect on carbohydrate and lipid metabolism | 6 hours postprandially

SECONDARY OUTCOMES:
Postprandial concentrations of glucose, non esterified fatty acids, insulin and triglycerides | 6 hours postprandially
Carbohydrate and lipid oxidation | 6 hours postprandially

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche En Nutrition Humaine Rhone Alpes, Lyon, France